CLINICAL TRIAL: NCT01952782
Title: Neuropeptides in Human Reproduction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013P001543
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Reproductive disorders; Hypogonadotropic hypogonadism; Kisspeptin; GnRH; Naloxone
MeSH Terms: conditions — Hypogonadism | interventions — Naloxone; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Naloxone, Kisspeptin, GnRH (Experimental): Intravenous (IV) administration of kisspeptin 112-121, GnRH, and naloxone
  Interventions: Drug: Kisspeptin 112-121; Drug: Naloxone; Drug: GnRH

INTERVENTIONS:
Drug: Kisspeptin 112-121 — Subjects will receive up to 10 IV doses of kisspeptin 112-121
  Other Names: Metastin 45-54
Drug: Naloxone — Subjects will receive one IV dose of naloxone followed by an IV infusion of naloxone.
Drug: GnRH — Subjects will receive up to 10 doses of IV GnRH
  Other Names: Gonadotropin-releasing hormone

SUMMARY:
The investigators are seeking healthy volunteers and volunteers with reproductive disorders for the study of the role of dynorphin in the reproductive system. Dynorphin is a naturally occurring opioid hormone that is blocked by naloxone.

We hypothesize that naloxone, by blocking dynorphin, will stimulate production of gonadotropin-releasing hormone (GnRH) and kisspeptin, two other naturally occurring reproductive hormones.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-40 (healthy men and regularly cycling women) OR ages 18-75 (men and women with hypogonadotropic hypogonadism (HH))
* Normal blood pressure (systolic BP <140 mm Hg, diastolic BP <90 mm Hg)
* White blood cell, platelets, prolactin, and thyroid stimulating hormone (TSH)within 90%-110% of laboratory reference range
* Negative urine drug screen panel
* Hemoglobin:

  1. For healthy men and healthy regularly cycling women: normal
  2. For men and women with HH: No less than 0.5 gm/dL below the lower limit of the reference range for normal women
* Blood urea nitrogen (BUN), creatinine, liver function tests not elevated
* For healthy subjects: Normal reproductive function and history
* For healthy subjects: Body Mass Index (BMI) 18.5-30kg/m2
* For subjects with HH: All medical conditions stable and well controlled

Exclusion Criteria:

* History of medication reaction requiring emergency medical attention
* Illicit drug use
* Consumption of more than 10 alcoholic drinks per week
* Difficulty with blood draws
* Currently seeking fertility, breastfeeding, or pregnant
* For healthy subjects: history of chronic disease and prescription medication use (with the exception of seasonal allergy medication)
* For subjects with HH: prescription medications known to affect reproductive endocrine function except for those used to treat the subject's reproductive condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Average difference in luteinizing hormone (LH) concentration before and after kisspeptin | Within 30 minutes of administration
  Compares response to kisspeptin on and off naloxone infusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lippincott MF, Leon S, Chan YM, Fergani C, Talbi R, Farooqi IS, Jones CM, Arlt W, Stewart SE, Cole TR, Terasawa E, Hall JE, Shaw ND, Navarro VM, Seminara SB. Hypothalamic Reproductive Endocrine Pulse Generator Activity Independent of Neurokinin B and Dynorphin Signaling. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4304-4318. doi: 10.1210/jc.2019-00146. PMID 31132118
- [Derived] Chan YM, Lippincott MF, Kusa TO, Seminara SB. Divergent responses to kisspeptin in children with delayed puberty. JCI Insight. 2018 Apr 19;3(8):e99109. doi: 10.1172/jci.insight.99109. eCollection 2018 Apr 19. PMID 29669934